CLINICAL TRIAL: NCT00047463
Title: Effects of Treating Obstructive Sleep Apnea in Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Beth Ann Malow, Professor of Neurology, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB030633; 1R01NS042698-01A1 (NIH)
Record Dates: First submitted 2002-10-07; First posted 2002-10-08 (Estimated); Results first posted 2011-05-03 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Epilepsy; Sleep Apnea; Obstructive Sleep Apnea
Keywords: epilepsy; sleep apnea; obstructive sleep apnea; continuous positive airway pressure; CPAP
MeSH Terms: conditions — Epilepsy; Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP active comparator (Active Comparator): continuous positive airway pressure (CPAP)
  Interventions: Device: continuous positive airway pressure (CPAP)
- CPAP Placebo (Placebo Comparator): Placebo-CPAP
  Interventions: Device: Placebo-CPAP

INTERVENTIONS:
Device: continuous positive airway pressure (CPAP) — a mask treatment for sleep apnea
  Arms: CPAP active comparator
Device: Placebo-CPAP — Placebo-CPAP
  Arms: CPAP Placebo

SUMMARY:
The purpose of this trial is to work out design issues prior to conducting a definitive phase 3 trial to determine whether treating sleep-related breathing disorders in people with epilepsy results in improvement in seizure control or an improvement in alertness during the day.

DETAILED DESCRIPTION:
Despite appropriate treatment with medications, individuals with epilepsy often continue to have seizures, and many suffer from excessive daytime sleepiness and poor quality of life. Evidence from case studies suggests that treatment of coexisting obstructive sleep apnea (OSA)-stoppage in breathing during sleep-can reduce the frequency of seizures in people with epilepsy that is resistant to antiepileptic medication.

In this study, individuals with symptoms of OSA and 2 or more seizures a month who meet study criteria will undergo polysomnography, a test that continuously monitors normal and abnormal physiological activity during sleep. Those individuals who test positive for OSA will be randomized to either therapeutic or placebo continuous positive airway pressure (CPAP)-a mask treatment for sleep apnea-for 10 weeks, during which time seizure frequency, daytime sleepiness, health-related quality of life, and CPAP compliance will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older.
* A history supportive of obstructive sleep apnea.
* Subject is able and willing to provide informed consent and to cooperate with polysomnography.
* Four or more quantifiable seizures per month.
* Subjects and their physicians agree to have their medication regimens optimized so that they are on the best regimen titrated to therapeutic benefit prior to the baseline phase of the study.

Exclusion Criteria:

* Seizures secondary to drugs, alcohol, infection, neoplasia, demyelination, metabolic illness, or progressive degenerative disease.
* Non-epileptic spells (e.g., pseudoseizures) alone or in combination with epileptic seizures.
* Narcolepsy or another primary sleep disorder that requires intervention with medications and which may affect results of study (e.g., severe periodic limb movement disorder).
* Effectively treated OSA or prior exposure to continuous positive airway pressure.
* History of poor compliance with antiepileptic medications.
* Current treatment with the vagus nerve stimulator.
* Pregnancy.
* A significant history of medical or psychiatric disease which may impair participation in the trial.
* A history of alcohol or drug abuse during the one-year period prior to trial participation.
* Evidence of medical instability (e.g., congestive heart failure, cardiac arrhythmias, pulmonary disease) due to obstructive sleep apnea.
* Subjects who are unaware of the majority of their seizures and lack a reliable witness.
* Greater than ten seizures a day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2002-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Malow, M.D., M.S., Principal Investigator — Vanderbilt University
Locations (4):
- United States (4):
  - University of Michigan, Ann Arbor, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Result] Malow BA, Foldvary-Schaefer N, Vaughn BV, Selwa LM, Chervin RD, Weatherwax KJ, Wang L, Song Y. Treating obstructive sleep apnea in adults with epilepsy: a randomized pilot trial. Neurology. 2008 Aug 19;71(8):572-7. doi: 10.1212/01.wnl.0000323927.13250.54. PMID 18711110
- [Result] Selwa LM, Marzec ML, Chervin RD, Weatherwax KJ, Vaughn BV, Foldvary-Schaefer N, Wang L, Song Y, Malow BA. Sleep staging and respiratory events in refractory epilepsy patients: Is there a first night effect? Epilepsia. 2008 Dec;49(12):2063-8. doi: 10.1111/j.1528-1167.2008.01681.x. Epub 2008 May 29. PMID 18513353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This pilot clinical trial was conducted between September 2002 and July 2005 at University of Michigan, Cleveland Clinic, University of North Carolina at Chapel Hill, and Vanderbilt University, with a Data Coordinating Center at the University of Michigan. 68 participants were enrolled and 35 were randomized.
Pre-assignment Details: Epilepsy clinic patients initially meeting trial eligibility on the basis of chart review completed a validated instrument that assesses the likelihood of having obstructive sleep apnea, and underwent a sleep and epilepsy evaluation by the site investigator. 68 patients consented, 33 not randomized due to not meeting criteria or declined.
Groups:
- Placebo Continuous Positive Airway Pressure: With placebo continuous positive airway pressure, the subject feels like he/she is receiving the real treatment because of the presence of a blower and mask. However, there is a large leak that prevents the subject from receiving adequate pressurized air to keep the airway open.
- Continuous Positive Airway Pressure: Continuous positive airway pressure is a standard treatment for obstructive sleep apnea that uses pressurized air delivered through a mask to keep the airway open and prevent obstruction during sleep.
Period: Overall Study
Arm/Group | Placebo Continuous Positive Airway Pressure | Continuous Positive Airway Pressure
Started | 13 | 22
Completed | 13 | 19
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Continuous Positive Airway Pressure | Continuous Positive Airway Pressure | Total
Number analyzed (Participants) | 13 | 22 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 22 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (14.3) | 42.7 (12.3) | 41.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 6 | 14 | 20
Region of Enrollment [Number; unit: participants]
  United States | 13 | 22 | 35

OUTCOME MEASURES:

1. Primary Outcome: CPAP Adherence/Tolerance as Measured by Proportion of Nights Used
Description: This measure quantifies how well patients use their CPAP. The standard unit of measurement is proportion of nights that the CPAP is used by a participant (total nights used/total nights the device could have been used), averaged across all participants . Data were downloaded by a card placed in the CPAP machine reflecting use over the entire 10 weeks.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: proportion of nights used (total nights
Arm/Group | Placebo Continuous Positive Airway Pressure | Continuous Positive Airway Pressure
Number analyzed (Participants) | 13 | 22
proportion of nights used (total nights | 0.74 (0.24) | 0.66 (0.3)
Statistical Analysis 1: Comparison: Placebo Continuous Positive Airway Pressure vs Continuous Positive Airway Pressure; The null hypothesis was that the groups would be similar in tolerance. This was a pilot study so we did not do a power calculation; Test type: Superiority or Other; p = 0.26, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Patients That Were Able to be Blinded to CPAP or Placebo CPAP
Description: Patients all received a CPAP machine which either delivered CPAP or provided the patient with placebo CPAP, which had the same sensation as receiving CPAP
Time Frame: 10 weeks
Measure: Number; unit: participants
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Placebo-CPAP
Number analyzed (Participants) | 22 | 13
participants | 22 | 13

3. Secondary Outcome: Number of Patients Requiring Only One Night of Baseline Sleep Study to Detect Sleep Apnea
Description: The data presented below represent the number of participants who required only one night of baseline sleep study prior to randomization
Time Frame: prior to randomization
Population: These are participants that were enrolled and assessed to determine if one night of baseline sleep study was sufficient to detect sleep apnea. This occurred prior to randomization. Five of the assessed participants were not randomized.
Measure: Number; unit: Participants
Arm/Group | All Participants Prior to Randomization
Number analyzed (Participants) | 40
Participants | 39

ADVERSE EVENTS:
Arm/Group | Placebo Continuous Positive Airway Pressure | Continuous Positive Airway Pressure
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/22
Other Adverse Events (participants affected / at risk) | 2/13 | 5/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Continuous Positive Airway Pressure (N=13) | Continuous Positive Airway Pressure (N=22)
tachycardia or chest tightness (Cardiac disorders) | 1 (1) | 1 (1) — patient described a rapid heart rate
skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) — Skin irritation at site of CPAP mask
nasal congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) — nasal congestion for CPAP use
GI discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) — Gastrointestinal discomfort after use of CPAP
anxiety (Psychiatric disorders) | 1 (1) | 0 (0) — anxious using CPAP

LIMITATIONS AND CAVEATS:
Being a pilot study with a relatively small sample size, we were unable to isolate the effects of specific medications or seizure types on the presence of sleep apnea.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No